CLINICAL TRIAL: NCT01132664
Title: A Phase Ib/II, Open Label, Multi-center Study Evaluating the Safety and Efficacy of BKM120 in Combination With Trastuzumab in Patients With Relapsing HER2 Overexpressing Breast Cancer Who Have Previously Failed Trastuzumab
Brief Title: Phase 1b/2 Study of BKM120 Plus Trastuzumab in Patients With HER2-positive Breast Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to the rare patient population and challenges to enroll patients.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBKM120X2107; 2009-015417-46 (EudraCT Number)
Record Dates: First submitted 2010-05-07; First posted 2010-05-28 (Estimated); Results first posted 2015-10-30 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Metastatic Breast Cancer; HER2+ Breast Cancer
Keywords: HER2; BKM120; PIK3; metastatic breast cancer; brain metastases; Herceptin; trastuzumab; capecitabine; open-label; maximum tolerated dose; Phase I/Phase ll
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms | interventions — NVP-BKM120; Trastuzumab; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HER2+ metastatic breast cancer (Experimental): Patients with HER2-overexpressing metastatic breast cancer, with or without PIK3 signaling pathway alteration, who have previously failed trastuzumab
  Interventions: Drug: BKM120; Drug: Trastuzumab
- HER2+ metastatic breast cancer with BM (Experimental): Patients with HER2-overexpressing metastatic breast cancer and brain metastases, with or without PIK3 signaling pathway alteration, who have previously failed trastuzumab
  Interventions: Drug: BKM120; Drug: Trastuzumab; Drug: Capecitabine

INTERVENTIONS:
Drug: BKM120 — Buparlisib (BKM120) is the investigational drug. Burparlisib was supplied as 10 mg and 50 mg hard gelatin capsules. Buparlisib was dosed on a flat scale of mg/day and not adjusted to body weight or body surface area. Buparlisib capsules were packaged in high density polyethylene bottles with a plastic child resistant closure.
Drug: Trastuzumab — Trastuzumab was used in this study according to the local regulations in each participating country. A loading dose (4 mg/kg) of trastuzumab was administered (if required as assessed by the principal Investigator based on the timing of the last trastuzumab dose prior to enrollment) on Day -7 over 90 minutes, followed by weekly intravenous infusion of 2 mg/kg maintenance doses from Day 1 of Cycle 1 (over 30 minutes if the previous infusion was well tolerated).
Drug: Capecitabine — 1000 mg/m2 twice a day from day 1 to Day 14 of a 21-day cycle.
  Arms: HER2+ metastatic breast cancer with BM

SUMMARY:
This study will assess the safety and efficacy of BKM120 in combination with trastuzumab in patients with relapsing HER2 overexpressing breast cancer who have previously failed trastuzumab.

The study will further assess the safety and preliminary efficacy of BKM120 in combination with trastuzumab and capecitabine in patients with relapsing HER2 overexpressing breast cancer and brain metastases (BM) who have previously failed trastuzumab.

ELIGIBILITY:
Inclusion Criteria:

* World Health Organization (WHO) Performance Status of ≤ 2
* Patients with HER2+ breast cancer by local laboratory testing (immunohistochemistry [IHC] 3+ staining or fluorescence in situ hybridization [FISH] confirmation for IHC 2+ and 1+)
* Documented tumor resistance to trastuzumab:

  * Recurrence while on trastuzumab or within 12 months since the last infusion for patients who received trastuzumab as adjuvant treatment
  * Progression while on or within 4 weeks since the last infusion of trastuzumab for patients who received trastuzumab for metastatic disease.
* Documented evidence of progressive disease per Response Evaluation Criteria in Solid Tumors (RECIST) on trastuzumab-based therapy defined as:

  * Phase Ib: at any time before study entry
  * Phase II: within 16 weeks before date of first dosing
* Received at least 1 but no more than 4 prior anit-HER2 based regimens including at least 1 regimen containing trastuzumab (adjuvant or neo-adjuvant trastuzumab will be considered as one prior regimen). HER2 directed therapies are defined as comprising trastuzumab, lapatinib, and trastuzumab-DM1 (T-DM1) only.

  • Phase II only: trastuzumab, T-DM1 or lapatinib must be part of the most recent line of therapy
* Previous lines of cytotoxic chemotherapy:

  * Phase Ib: no more than 4 lines of cytotoxic chemotherapy
  * Phase II: no more than 3 lines of cytotoxic chemotherapy

Measurable disease:

* Phase Ib: patient has at least one measurable lesion or non-measurable disease as defined per RECIST
* Phase II: patient has at least one measureable lesion as defined per RECIST

|| Specific Inclusion Criteria for patients in BM cohorts:

* Patient has evidence of progressing brain metastases and/or new metastatic brain lesion(s) without leptomeningeal disease.
* Patient has received prior WBRT and/or SRS at at >28 and >/= 14 days, respectively, prior to starting study drug and the patient must have recovered from the side effects of the therapy
* WHO performance status of </=1
* PT INR </= 1.5
* Any number of prior HER2-directed and cytotoxic regimens, and the most recent line may be any type of anti-neoplastic therapy

|| Exclusion Criteria:

* Patients with untreated brain metastases
* Patients with acute or chronic liver, renal disease or pancreatitis
* Patients with any peripheral neuropathy ≥ Common Terminology Criteria for Adverse Events (CTCAE) grade 2
* Patients with a history of mood disorders or ≥ CTCAE grade 3 anxiety
* Patient with clinical manifest diabetes mellitus or steroid-induced diabetes mellitus

|| Specific Exclusion Criteria for patients in BM cohorts

* Prior treatment with capecitabine
* Patient has known dihydropyrimidine dehydrogenase (DPD) deficiency
* Patient is currently receiving treatment with EIAED
* Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2010-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (21):
- United States (7):
  - University of Alabama at Birmingham/ Kirklin Clinic Univ AL - PI, Birmingham, Alabama
  - Highlands Oncology Group Dept of Highlands Oncology Grp, Fayetteville, Arkansas
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Karmanos Cancer Institute Dept.of KarmanosCancerInst (6), Detroit, Michigan
  - Washington University School Of Medicine-Siteman Cancer Ctr WA Siteman, St Louis, Missouri
  - Beth Israel Medical Center BIMC, New York, New York
  - Sarah Cannon Research Institute Sarah Cannon Cancer Center SC, Nashville, Tennessee
- Belgium (2):
  - Novartis Investigative Site, Liège
  - Novartis Investigative Site, Wilrijk
- France (2):
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Saint-Herblain Cédex
- Italy (4):
  - Novartis Investigative Site, Cagliari, CA
  - Novartis Investigative Site, Macerata, MC
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Terni, TR
- Spain (3):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, Valencia, Valencia
- United Kingdom (3):
  - Novartis Investigative Site, Brighton, East Sussex
  - Novartis Investigative Site, Nottingham
  - Novartis Investigative Site, Oxford

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 72 patients (pts) were enrolled: 18 in ph lb, 53 in ph ll, including 8 from ph lb, with 45 new pts in ph ll & 9 in the brain metastasis (BM) cohort. Of the 72 pts, 1 in ph lb & 3 in phase ll, did not receive Burparlisib, only Trastuzumab. Therefore, 68 patients (17 in ph l, 42 in ph ll, 9 in BM cohort) were treated with buparlisib + trastuzumab.
Pre-assignment Details: Primary outcome measure for BM cohort was MTD/RP2D which was not reached/established due to premature termination of the study.
  Objective Response Rate (ORR), Disease Control Rate (DCR), Clinical Benefit Rate (CBR) & Progression Free Survival (PFS)were not calculated for the BM cohort either.
Groups:
- Phase Ib - 50 mg: Patients in the phase Ib dose escalation cohort who received 50 mg of buparlisib - investigational drug
- Phase Ib - 100mg: Patients in the phase Ib dose escalation cohort who received 100 mg of buparlisib - investigational drug
- Phase II - 100mg: Patients in the phase II expansion + patients from phase Ib dose escalation were included in phase II and received 100 mg of investigational drug - buparsilib
- BM Cohort - 80mg: Patients in the BM cohort who received 80 mg of buparlisib - investigational drug
- BM Cohort - 100mg: Patients in the BM cohort who received 100 mg of buparlisib - investigational drug
Period: Phase lb
Arm/Group | Phase Ib - 50 mg | Phase Ib - 100mg | Phase II - 100mg | BM Cohort - 80mg | BM Cohort - 100mg
Started | 5 | 12 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 5 | 12 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 0 | 0
Not completed — Disease Progression | 4 | 9 | 0 | 0 | 0
Period: Phase ll
Arm/Group | Phase Ib - 50 mg | Phase Ib - 100mg | Phase II - 100mg | BM Cohort - 80mg | BM Cohort - 100mg
Started | 0 | 0 | 50 (Of the 50 patients, 8 were from phase lb & were eligible for inclusion in Phase II) | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 50 | 0 | 0
Not completed — Death | 0 | 0 | 2 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 10 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 0 | 0
Not completed — Disease progression | 0 | 0 | 35 | 0 | 0
Period: BM Cohort
Arm/Group | Phase Ib - 50 mg | Phase Ib - 100mg | Phase II - 100mg | BM Cohort - 80mg | BM Cohort - 100mg
Started | 0 | 0 | 0 | 3 | 6
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 3 | 6
Not completed — Disease progression | 0 | 0 | 0 | 3 | 4
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Phase II - 100mg: Patients in the phase II only expansion cohort who received 100 mg of buparlisib - investigational drug
- Total: Total of all reporting groups
Arm/Group | Phase Ib - 50 mg | Phase Ib - 100mg | Phase II - 100mg | BM Cohort - 80mg | BM Cohort - 100mg | Total
Number analyzed (Participants) | 5 | 12 | 42 | 3 | 6 | 68
Age, Customized [Number; unit: Participants]
  <65 years | 5 | 11 | 35 | 3 | 6 | 60
  >=65 years | 0 | 1 | 7 | 0 | 0 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 12 | 42 | 3 | 6 | 68
  Male | 0 | 0 | 0 | 0 | 0 | 0
Female: Child bearing potential [Number; unit: Participants]
  Able to bear children | 2 | 3 | 8 | 1 | 1 | 15
  Premenarche | 0 | 0 | 0 | 0 | 0 | 0
  Post-menopausal | 3 | 8 | 31 | 2 | 4 | 48
  Sterile - of child bearing age | 0 | 1 | 3 | 0 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicity (DLT) - Phase l Only
Description: Determination of the maximum tolerated dose (MTD) in the dose escalation part of the study was based upon the estimation of the probability of DLT in Cycle 1 in patients of the dose-determining set.
Time Frame: cycle 1 - 28 days
Population: The Dose-determining set (DDS) for the determination of the MTD consisted of all patients from the safety set in the dose escalation phase who had met the minimum safety evaluation requirements and the minimum exposure criterion or had experienced DLT during Cycle 1 and were discontinued. MTD analysis was done only on the phase lb group.
Measure: Number; unit: Participants
Groups:
- Phase II - 100mg: Patients in the phase II expansion + patients from phase Ib escalation included in phase II
Arm/Group | Phase Ib - 50 mg | Phase Ib - 100mg | Phase II - 100mg | BM Cohort - 80mg | BM Cohort - 100mg
Number analyzed (Participants) | 4 | 11 | 0 | 3 | 5
Participants
  Primary system orgran class (SOC) PT - grade 1 | 0 | 0 |  | 0 | 0
  Primary SOC PT - grade 2 | 0 | 0 |  | 0 | 0
  Primary SOC PT (asthenia) - grade 3 | 0 | 1 |  | 0 | 0
  Primary SOC PT - grade 4 | 0 | 0 |  | 0 | 0
  Primary SOC PT - missing | 0 | 0 |  | 0 | 0
  Primary SOC PT (somatits/diarrhea) - grade 3 | 0 | 0 |  | 0 | 1

2. Primary Outcome: Overall Response Rate (ORR) - Phase ll
Description: Objective response rate (ORR) was defined as the rate of patients with best overall response (BOR) equal to complete response (CR) or partial response (PR) according to RECIST 1.0 from the Investigators review.
  Per Response Evaluation Criteria In Solid Tumors (RECIST) version 1.0 assessed of the disease status by imaging (i.e. CT/MRI): Complete Response (CR) = Disappearance of all tumor lesions; Partial Response (PR)= >=30% shrinkage of lesions; Overall Response (OR) = patients with CR and PR.
Time Frame: 18 months
Population: The full analysis set (FAS) consisted of all patients who received at least one dose of study drug (buparlisib)
Measure: Number; unit: Participants
Arm/Group | Phase Ib - 50 mg | Phase Ib - 100mg | Phase II - 100mg | BM Cohort - 80mg | BM Cohort - 100mg
Number analyzed (Participants) | 0 | 0 | 50 | 0 | 0
Participants |  |  | 5 |  |

3. Secondary Outcome: Disease Control Rate (DCR) Based on Investigator Assessment- Phase l & ll
Description: Disease control rate (DCR) = patients with complete response (CR), partial response (PR) or stable disease (SD) as per RECIST criteria.
  Response Evaluation Criteria In Solid Tumors (RECIST) version 1.0 assessed the disease status by imaging (i.e. CT/MRI): CR = disappearance of all tumor lesions; PR = >=30% shrinkage of lesions; SD = Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progressive disease (PD); PD = At least a 20% increase in the sum of the longest diameter of all measured target lesions, taking as reference the smallest sum of longest diameter of all target lesions recorded at or after baseline.
Time Frame: 18 months
Population: The full analysis set (FAS) consisted of all patients who received at least one dose of study drug (buparlisib).
  CBR analysis was not done for the BM cohort population. DCR analysis was not done for the BM cohort population.
Measure: Number; unit: Participants
Arm/Group | Phase Ib - 50 mg | Phase Ib - 100mg | Phase II - 100mg | BM Cohort - 80mg | BM Cohort - 100mg
Number analyzed (Participants) | 5 | 12 | 50 | 0 | 0
Participants
  Phase l | 1 | 7 | 0 |  |
  Phase ll | 0 | 0 | 25 |  |

4. Secondary Outcome: Clinical Benefit Rate (CBR) - Phase l & ll
Description: CBR = patients with CR, PR or SD ≥ 24 weeks according to RECIST by the investigator.
  Response Evaluation Criteria In Solid Tumors (RECIST) version 1.0 assessed the disease status by imaging (i.e. CT/MRI): CR = Disappearance of all tumor lesions; PR= >=30% shrinkage of lesions; SD = Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for PD; PD = At least a 20% increase in the sum of the longest diameter of all measured target lesions, taking as reference the smallest sum of longest diameter of all target lesions recorded at or after baseline.
Time Frame: 18 months
Population: The full analysis set (FAS) consisted of all patients who received at least one dose of study drug (buparlisib).
  CBR analysis was not done for the BM cohort population.
Measure: Number; unit: Participants
Arm/Group | Phase Ib - 50 mg | Phase Ib - 100mg | Phase II - 100mg | BM Cohort - 80mg | BM Cohort - 100mg
Number analyzed (Participants) | 5 | 12 | 50 | 0 | 0
Participants
  Phase l | 0 | 3 | 0 |  |
  Phase ll | 0 | 0 | 7 |  |

5. Secondary Outcome: Progression Free Survival (PFS) - Based on Investigator Review Using Kaplan Meier - Phase l & ll
Time Frame: 18 months
Population: FAS consisted of all patients who received at least 1 dose of study drug (buparlisib). PFS analysis was not done for the BM cohort population. MTD/RP2D was not established due to premature termination of the study. In the phase ll portion of the study, PFS was analyzed only in patients with known PIK3 status, thus only 26/50 patients were analyzed.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Phase Ib - 50 mg | Phase Ib - 100mg | Phase II - 100mg | BM Cohort - 80mg | BM Cohort - 100mg
Number analyzed (Participants) | 5 | 12 | 26 | 0 | 0
Months
  Phase l | 1.7 [1.3 to 3.6] | 3.3 [1.6 to 5.4] | NA [NA to NA] — NA = data reported here for phase l only and not for phase ll |  |
  Phase ll: PIK3CA wildtype (n =18) | NA [NA to NA] — NA = data reported here for phase ll only and not for phase l | NA [NA to NA] — NA = data reported here for phase ll only and not for phase l | 1.7 [1.5 to 5.4] |  |
  Phase ll: PIK3CA mutated (n =8) | NA [NA to NA] — NA = data reported here for phase ll only and not for phase l | NA [NA to NA] — NA = data reported here for phase ll only and not for phase l | 1.8 [1.3 to 3.4] |  |

ADVERSE EVENTS:
Groups:
- Phase Ib Dose Escalation 50 mg/Day: Patients in the phase Ib dose escalation cohort who received 50 mg of buparlisib - investigational drug.
- Phase Ib Dose Escalation 100 mg/Day: Patients in the phase Ib dose escalation cohort who received 100 mg of buparlisib - investigational drug
- Phase II Dose Expansion 100 mg/Day: Patients in the phase II expansion + patients from phase Ib dose escalation who received 100 mg/day of buparlisib - investigational drug
- BM Cohort 80 mg/Day: Patients in the BM cohort who received 80 mg of buparlisib - investigational drug
- BM Cohort 100 mg/Day: Patients in the BM cohort who received 100 mg of buparlisib - investigational drug
Arm/Group | Phase Ib Dose Escalation 50 mg/Day | Phase Ib Dose Escalation 100 mg/Day | Phase II Dose Expansion 100 mg/Day | BM Cohort 80 mg/Day | BM Cohort 100 mg/Day
Serious Adverse Events (participants affected / at risk) | 2/5 | 2/12 | 17/50 | 2/3 | 4/6
Other Adverse Events (participants affected / at risk) | 5/5 | 12/12 | 50/50 | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase Ib Dose Escalation 50 mg/Day (N=5) | Phase Ib Dose Escalation 100 mg/Day (N=12) | Phase II Dose Expansion 100 mg/Day (N=50) | BM Cohort 80 mg/Day (N=3) | BM Cohort 100 mg/Day (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 3 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Asthenia (General disorders) | 0 | 2 | 3 | 0 | 0
General Physical Health Deterioration (General disorders) | 0 | 0 | 1 | 0 | 0
Oedema Peripheral (General disorders) | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0 | 0
Systemic Inflammatory Response Syndrome (General disorders) | 0 | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Hepatic Failure (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1
Device Related Infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Lobar Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Lung Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 2 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 1 | 0 | 0
Bilirubin Conjugated Increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood Bilirubin Increased (Investigations) | 0 | 0 | 1 | 0 | 0
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Cerebral Haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Status Epilepticus (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Affective Disorder (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0
Confusional State (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Depressed Mood (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Mood Altered (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase Ib Dose Escalation 50 mg/Day (N=5) | Phase Ib Dose Escalation 100 mg/Day (N=12) | Phase II Dose Expansion 100 mg/Day (N=50) | BM Cohort 80 mg/Day (N=3) | BM Cohort 100 mg/Day (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 5 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 3 | 1 | 0
Dry Eye (Eye disorders) | 0 | 2 | 2 | 0 | 0
Extraocular Muscle Paresis (Eye disorders) | 0 | 1 | 1 | 0 | 0
Eye Irritation (Eye disorders) | 0 | 0 | 0 | 1 | 0
Eye Pain (Eye disorders) | 0 | 0 | 0 | 1 | 0
Ocular Hyperaemia (Eye disorders) | 0 | 0 | 0 | 1 | 0
Photophobia (Eye disorders) | 0 | 1 | 1 | 0 | 0
Vision Blurred (Eye disorders) | 0 | 1 | 1 | 2 | 1
Visual Impairment (Eye disorders) | 1 | 0 | 1 | 1 | 1
Abdominal Distension (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 3 | 7 | 0 | 1
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 2 | 5 | 1 | 1
Anal Fissure (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Aphthous Stomatitis (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 6 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 5 | 25 | 3 | 5
Dry Mouth (Gastrointestinal disorders) | 0 | 1 | 2 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 6 | 3 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 3 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Haemorrhoids Thrombosed (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Lip Ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Mouth Ulceration (Gastrointestinal disorders) | 0 | 1 | 3 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 24 | 2 | 4
Pigmentation Lip (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 4 | 12 | 1 | 2
Tongue Discolouration (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Tooth Disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2 | 13 | 1 | 4
Asthenia (General disorders) | 1 | 6 | 13 | 0 | 1
Chest Pain (General disorders) | 0 | 1 | 1 | 0 | 0
Face Oedema (General disorders) | 0 | 0 | 1 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 16 | 3 | 4
Gait Disturbance (General disorders) | 0 | 0 | 0 | 1 | 0
Injection Site Reaction (General disorders) | 0 | 0 | 0 | 1 | 0
Mucosal Dryness (General disorders) | 0 | 2 | 1 | 0 | 0
Mucosal Inflammation (General disorders) | 0 | 0 | 0 | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 7 | 1 | 0
Oedema Peripheral (General disorders) | 0 | 0 | 3 | 0 | 0
Pain (General disorders) | 0 | 1 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 5 | 1 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Device Related Sepsis (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Ear Infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Eczema Infected (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Furuncle (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Herpes Zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 0 | 2 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Oral Herpes (Infections and infestations) | 0 | 0 | 3 | 0 | 0
Paronychia (Infections and infestations) | 0 | 1 | 2 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 1 | 2 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Spinal Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
Tooth Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Vaginal Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Wound Complication (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Alanine Aminotransferase Decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 1 | 4 | 18 | 0 | 1
Amylase Increased (Investigations) | 0 | 1 | 1 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 1 | 4 | 17 | 0 | 1
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 2 | 7 | 0 | 0
Blood Bilirubin Increased (Investigations) | 0 | 0 | 3 | 0 | 0
Blood Calcium Decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood Cholesterol Increased (Investigations) | 0 | 1 | 1 | 0 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 0 | 0 | 1 | 1 | 0
Blood Creatinine Increased (Investigations) | 0 | 1 | 2 | 0 | 0
Blood Glucose Decreased (Investigations) | 0 | 1 | 1 | 0 | 0
Blood Glucose Increased (Investigations) | 0 | 1 | 2 | 0 | 0
Blood Thyroid Stimulating Hormone Increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood Uric Acid Increased (Investigations) | 0 | 1 | 1 | 0 | 0
C-Reactive Protein Increased (Investigations) | 0 | 0 | 1 | 1 | 0
Eastern Cooperative Oncology Group Performance Status Worsened (Investigations) | 0 | 1 | 3 | 0 | 0
Ejection Fraction Decreased (Investigations) | 0 | 1 | 2 | 0 | 0
Gamma-Glutamyltransferase Increased (Investigations) | 1 | 3 | 7 | 0 | 0
Glycosylated Haemoglobin Increased (Investigations) | 0 | 0 | 0 | 1 | 0
Haemoglobin Decreased (Investigations) | 1 | 0 | 1 | 0 | 0
Insulin C-Peptide Increased (Investigations) | 0 | 0 | 1 | 1 | 0
Lipase Increased (Investigations) | 0 | 1 | 1 | 0 | 1
Liver Function Test Abnormal (Investigations) | 0 | 0 | 1 | 0 | 1
Low Density Lipoprotein Increased (Investigations) | 1 | 0 | 0 | 0 | 0
Lymphocyte Count Decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Protein Urine Present (Investigations) | 0 | 1 | 1 | 0 | 0
Weight Decreased (Investigations) | 1 | 1 | 7 | 1 | 1
White Blood Cell Count Decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 1 | 18 | 2 | 4
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 5 | 15 | 1 | 1
Hyperphagia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 3 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 0 | 0
Increased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 6 | 0 | 2
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4 | 2 | 2
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 5 | 0 | 1
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0
Balance Disorder (Nervous system disorders) | 0 | 1 | 5 | 1 | 0
Cluster Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 6 | 1 | 1
Dysgeusia (Nervous system disorders) | 1 | 1 | 7 | 1 | 1
Headache (Nervous system disorders) | 1 | 1 | 11 | 1 | 2
Memory Impairment (Nervous system disorders) | 0 | 0 | 2 | 1 | 0
Neuropathy Peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 1 | 3 | 0 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 2 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Tremor (Nervous system disorders) | 1 | 0 | 3 | 1 | 1
Affective Disorder (Psychiatric disorders) | 0 | 3 | 5 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 11 | 1 | 2
Binge Eating (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Depressed Mood (Psychiatric disorders) | 0 | 0 | 3 | 0 | 0
Depression (Psychiatric disorders) | 2 | 1 | 8 | 0 | 1
Initial Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 2 | 6 | 1 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1
Mood Altered (Psychiatric disorders) | 3 | 4 | 7 | 0 | 1
Nervousness (Psychiatric disorders) | 0 | 1 | 1 | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Suicidal Ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0
Micturition Urgency (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Breast Pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 1
Vulvovaginal Discomfort (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 15 | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 6 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 4 | 1 | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Respiratory Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 3 | 6 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 3 | 0 | 0
Nail Disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1 | 3
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 3 | 7 | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 6 | 16 | 2 | 1
Rash Generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 0 | 0
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 4 | 0 | 0
Skin Discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Swelling Face (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 3 | 6 | 0 | 0
Orthostatic Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.